CLINICAL TRIAL: NCT06362005
Title: The Efficacy of Selenium as an Alternative or Complementary Topical Treatment of Oral Lichen Planus (Randomized Clinical Trial)
Brief Title: The Efficacy of Selenium as an Alternative or Complementary Topical Treatment of Oral Lichen Planus
Acronym: RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Sphinx university (Other)
Responsible Party: Principal Investigator, Shaymaa Hussein Rafat Kotb, Assistant lecturere of oral medicine ,periodontology departement, Sphinx university
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AUAREC2023011-1
Record Dates: First submitted 2024-03-27; First posted 2024-04-12 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Lichen Planus, Oral
Keywords: seleinum; Antioxidant; Glutathione-S-transferases; Reactive oxygen species
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Triamcinolone Acetonide; Ointments; Selenium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- group I (triamcinolone) (Placebo Comparator): ten patients with oral lichen planus, will receive topical triamcinolone acetonide 0.1% four times per day for six weeks.
  Interventions: Drug: Triamcinolone Acetonide 0.1% Oint
- group II (tacrollimus) (Placebo Comparator): ten patients with oral lichen planus, will receive topical tacrolimus 0.1% four times per day for six weeks.
  Interventions: Drug: Tacrollimus Topical
- group III (selenium) (Experimental): ten patients with oral lichen planus, will receive topical selenium four times per day for six weeks.
  Interventions: Drug: Selenium
- group IV (selenium + triamcinolone ) (Experimental): : ten patients with oral lichen planus, will receive topical selenium combined with topical triamcinolone acetonide 0.1% three times per day for each for six weeks
  Interventions: Drug: Selenium & Triamcinolone Acetonide 0.1% Oint
- group V ( selenium + tacrollimus) (Experimental): ten patients with oral lichen planus, will receive topical selenium combined with topical tacrolimus 0.1% three times per day for each for six weeks.
  Interventions: Drug: Selenium& Tacrollimus topical

INTERVENTIONS:
Drug: Triamcinolone Acetonide 0.1% Oint — RCT
  Other Names: Group I
  Arms: group I (triamcinolone)
Drug: Tacrollimus Topical — RCT
  Other Names: Group II
  Arms: group II (tacrollimus)
Drug: Selenium — RCT
  Other Names: Group III
  Arms: group III (selenium)
Drug: Selenium & Triamcinolone Acetonide 0.1% Oint — RCT
  Other Names: Group IV
  Arms: group IV (selenium + triamcinolone )
Drug: Selenium& Tacrollimus topical — RCT
  Other Names: Group V
  Arms: group V ( selenium + tacrollimus)

SUMMARY:
evaluate clinically and biochemically the efficacy of topically applied selenium as complementary or alternative to triamcinolone acetonide 0.1% and tacrolimus 0.1% in patients with oral lichen planus.

DETAILED DESCRIPTION:
The signs and symptoms of the oral lichen planus lesion. 2-The associated oral symptoms. 3- Glutathione biomarker level as an antioxidant enzyme in saliva by ELISA analysis .

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of OLP

Exclusion Criteria:

1. lichenoid reaction from medication ' .
2. any systemic autoimmune disease
3. Pregnancy
4. smokers

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
to assess a visual analog scale (VAS)of the oral lichen planus lesion | baseline, 1, 3 and 6 months after treatment
  qualitative

SECONDARY OUTCOMES:
to assess The associated Oral Disease Severity Score 3- Glutathione biomarker level as an antioxidant enzyme in saliva by ELISA analysis | baseline, 1, 3 and 6 months after treatment
  qualitative ,and quantitiave
Biochemical evaluation of salivary Glutathione level using (ELISA) | baseline, 1, 3 months after treatment
  Quantity

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar university ,faculty of Dental Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All patients were recruited from the outpatient clinic of the Dermatology Department, Assiut University Hospitals, and referred to oral Medicine clinics, Faculty of Dental Medicine, Al-Azhar University, Assiut branch.
Supporting Information: SAP
Time Frame: ready now

REFERENCES:
- See also: orcid — https://orcid.org/my-orcid?orcid=0000-0002-8404-438X
- See also: ncbi — https://www.ncbi.nlm.nih.gov/myncbi/shaymaa.kotb.1/cv/655768